CLINICAL TRIAL: NCT04328324
Title: Pattern of Upper Gastrointestinal Lesions in Upper Egypt : Clinical, Endoscopic and Pathological Evaluation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Radwa Hussein Mohammed Hasanen, RHMHasanen, Assiut University
Other Study IDs: 2832020
Record Dates: First submitted 2020-03-28; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Pattern of Upper Gastrointestinal Lesions
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopy — Diagnostic upper Git endoscopy

SUMMARY:
Upper Gastrointestinal (UGI) symptoms are among the commonest complaints for which patients seek medical attention, with the annual prevalence of dyspepsia approximating 25% . Endoscopy holds an important place in the diagnosis of UGI conditions by enabling visualization, photography, ultrasonography, and biopsying of suspicious lesions . It gives a better diagnostic yield over radiology particularly in the investigation of upper gastrointestinal bleeding, inflammatory conditions of the upper gastro-intestinal track like esophagitis, gastritis and duodenitis as well as the diagnosis of Mallory Weiss tears and vascular malformations .Dyspepsia in the absence of any other symptom was the indication for UGIE in the vast majority of patients. Close to 80% of our patients presented with dyspepsia not associated with any other symptom and in 50% of the patients the endoscopic findings were normal [4]. Other common reasons for UGIE were GERD symptoms, recurrent vomiting, dyspepsia associated with weight loss and patients with symptoms of UGI bleeding . Gastritis was the most frequent endoscopic finding in our patients, followed by duodenitis .Gastric ulcer was diagnosed more frequently than duodenal ulcers . Taking a biopsy is very helpful in diagnosis in our study. H. pylori colonization of the gut is the main cause of chronic gastritis and the principal etiological agent of gastric cancer and peptic ulcer disease . Gastric cancer was diagnosed, by endoscopy, about eight times more frequently in patients presenting with an alarm symptom like recurrent vomiting, dyspepsia together with weight loss or UGI bleeding .

ELIGIBILITY:
Inclusion Criteria:

- All patient undergoing elective and urgent upper GIT endoscopy either therapeutic or diagnostic.

Exclusion Criteria:

* Patient undergoing endoscopic intervention for previously detected endoscopic lesion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patient undergoing elective and urgent upper GIT endoscopy either therapeutic or diagnostic.
  In elrajhi endoscopy unit
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-30 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Pattern of upper gastrointestinal lesions | 1 year
  We will see what common GIT lesions happen in patients of upper Egypt

IPD SHARING:
Plan to Share IPD: Undecided